CLINICAL TRIAL: NCT02930161
Title: Многоцентровое двойное слепое плацебо-контролируемое рандомизированное исследование препарата Рунихол® у пациентов с неалкогольной жировой болезнью печени на фоне метаболического синдрома
Brief Title: Runihol in Nonalcoholic Fatty Liver Disease and Metabolic Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RUN-II-2015
Record Dates: First submitted 2016-10-06; First posted 2016-10-12 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Nonalcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis; Methionine; Succinic acid
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Runihol 2 tablets x 2 times a day (Experimental): Intake of 1 tablet of Runihol and 1 placebo tablet orally, with drinking 100 ml of water, 30 minutes before meals three times a day (morning, afternoon and evening) for 84 days (12 weeks).
  Interventions: Drug: Runihol
- Runihol 1 tablet x 3 times a day (Experimental): Intake of Runihol, 2 tablets orally, with drinking 100 ml of water, 30 minutes before meals, 2 times a day (morning and evening) for 84 days (12 weeks), and 2 placebo tablets orally, with drinking 100 ml of water, 30 minutes before meals, 1 time a day (afternoon) for 84 days (12 weeks).
  Interventions: Drug: Runihol
- Placebo (Placebo Comparator): Two placebo tablets orally, with drinking 100 ml of water, 30 minutes before meals three times a day (morning, afternoon and evening) for 84 days (12 weeks).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Runihol — Composition of Runihol®:
  One tablet contains:
  Active ingredients: succinic acid - 0.250 g; Riboxinum (inosine) - 0.100 g; taurine - 0.050 g; Methionine - 0.050 g Excipients - 0.184 g: potato starch, povidone, microcrystalline cellulose, calcium stearate, hypromellose, polysorbate-80.
  Enteric coat - 0.061 g: methacrylic acid-ethyl acrylate copolymer, talc, titanium dioxide, triethyl citrate, colloidal silicon dioxide, sodium hydrogencarbonate, sodium lauryl sulfate.
  Other Names: Runihol, coated pill, produced by POLYSAN Ltd (Russia)
  Arms: Runihol 1 tablet x 3 times a day; Runihol 2 tablets x 2 times a day
Other: Placebo — The composition of the drug in one tablet:
  Active substance: None. The tablet core - 0.634 g: potato starch, povidone, microcrystalline cellulose, calcium stearate, hypromellose, polysorbate-80.
  Enteric coat - 0.061 g: methacrylic acid-ethyl acrylate copolymer, talc, titanium dioxide, triethyl citrate, colloidal silicon dioxide, sodium hydrogencarbonate, sodium lauryl sulfate.
  Tablet weight enteric coated - 0.695 g
  Arms: Placebo

SUMMARY:
The study is designed to assess the safety and efficacy of different doses and dosing regimens of Runihol, tablets, enteric coated, produced by "NTFF" POLYSAN" (Russia), in prevention of liver disease progression in patients with non-alcoholic fatty liver disease and metabolic syndrome.

DETAILED DESCRIPTION:
The aim of this study is a comparative assessment of the safety and efficacy of different doses and dosing regimens of Runihol drug tablets, enteric coated, produced by "NTFF" POLYSAN "(Russia) and placebo tablets, enteric coated, produced by" NTFF "POLYSAN" (Russia), when administered to patients with non-alcoholic fatty liver disease and metabolic syndrome.

Design: a multicenter, prospective, randomized, double-blind, placebo-controlled comparative study in parallel groups.

The study will be performed on the outpatient basis under the supervision of the physician-researcher who will be in charge of screening and the whole course of study drug therapy.

The study consists of the following periods:

* Screening - preliminary examination of the eligible patients (duration 14 days).
* The period of therapy - the use of the study drug Runihol®, tablets, enteric coated, produced by "NTFF" POLYSAN "(Russian) or placebo tablets, enteric coated, produced by" NTFF "POLYSAN" LLC (Russia), during 84 days (12 weeks).

Following screening, patients who meet the inclusion criteria and have no criteria for exclusion will be randomly assigned into three study groups in the proportion of 1: 1: 1):

* Group I: treatment with Runihol®, 1 tablet 3 times a day, and placebo tablets, 1 tablet three times a day, for 84 days (12 weeks).
* Group II: treatment with Runihol®, 2 tablets 2 times a day, morning and evening, and placebo tablets, 2 tablets once a day, in the afternoon, for 84 days (12 weeks).
* Group III: patients will receive placebo tablets, 2 tablets 3 times a day, for 84 days (12 weeks).

Patient assessment will be carried out in the course of 6 visits.

Screening:

Visit 0 (-14 day ... Day 1) - Screening: preliminary evaluation of patients.

Period of treatment:

Visit 1 (Day 1) - evaluation of the patient based on the results of physical examination, assessment of vital signs, complex laboratory (clinical and biochemical blood tests, PTI, insulin resistance index calculation, the determination of homocysteine in the serum / plasma, general urine analysis) and instrumental (ECG ) investigations; randomization, the appointment of therapy, assessment of concomitant therapy, instructions to fill the patient's diary, registration of AEs.

Visit 2 (Day 15) - evaluation of the patient based on the results of physical examination, assessment of vital signs, laboratory complex (clinical and biochemical blood tests, PTI, determination of homocysteine in the blood serum, the total urine analysis) and instrumental (ECG) studies; control of intake of study medication / placebo, evaluation of concomitant therapy, checking patient diary, registration of AEs.

Visit 3 (Day 29) - evaluation of the patient based on the results of physical examination, assessment of vital signs, laboratory complex (clinical and biochemical blood tests, PTI, determination of homocysteine in the serum / plasma, total urine analysis) and instrumental (ECG ) investigations; control of intake of study medication / placebo, evaluation of concomitant therapy, checking patient diary, registration of AEs.

Visit 4 (Day 57) - evaluation of the patient based on the results of physical examination, assessment of vital signs, laboratory complex (clinical and biochemical blood tests, PTI, determination of homocysteine in the serum / plasma, total urine analysis) and instrumental (ECG ) studies; control of intake of study medication / placebo, evaluation of concomitant therapy, checking patient diary, registration of AEs.

Visit 5 (Day 85) - evaluation of the patient based on the results of physical examination, assessment of vital signs, laboratory complex (clinical and biochemical blood tests, PTI, determination of homocysteine in the serum / plasma, insulin resistance index calculation, the total urine analysis) and instrumental (ECG, ultrasound of the abdomen) investigations; control of intake of study medication / placebo, evaluation of concomitant therapy, checking patient diary, registration of AEs.

The study is expected to include, and randomize at least 162 patients (men and women aged 18 to 65 years) with clinically or histologically confirmed diagnosis of non-alcoholic fatty liver disease (code ICD-10: K76.0: Fatty degeneration of the liver, not classified elsewhere) in the form of non-alcoholic steatohepatitis and metabolic syndrome, provided with written informed consent to participate in the study, the relevant criteria for inclusion in the study and no criteria for exclusion; data collected will be used for further analysis of safety and efficacy .

In view of possible dropout of patients at screening and during the study a total of 204 patients are planned for inclusion.

ELIGIBILITY:
Inclusion Criteria:

1. A signed informed consent to participate in the study.
2. Men and women aged 18 to 65 years.
3. Diagnosis: non-alcoholic fatty liver disease (code ICD-10: K76.0 Fatty degeneration of the liver, not classified elsewhere), defined as non-alcoholic steatohepatitis.
4. Metabolic syndrome (according to the national criteria accepted in 2013).
5. The body mass index (BMI) of 30-45 kg / m2.
6. The presence of signs of steatosis on ultrasound examination of the liver (distal signal attenuation and / or increased echogenicity of the liver).
7. The level of total cholesterol> 6.0 mmol/l and / or triglyceride levels> 1.7 mmol/l.
8. ALT, AST serum levels exceed upper normal limits by 1,5-7 times.
9. GGT level higher that upper normal limit by 1,5-7 times.
10. The level of SBP>140 and / or DBP> 90 mm Hg or antihypertensive therapy required to maintain normal blood pressure values.
11. A negativepregnancy test for female participants.
12. Consent to use of appropriate methods of contraception ( with contraceptive reliability over 90%: the cervical cap with spermicide, diaphragm with spermicide, condoms, intrauterine devices), or abstaining from sexual activity for the study period.
13. Consent to limit alcohol consumption to a maximum of 2 units of alcohol per month (1 unit of alcohol is equivalent to 0.5 liters of beer, 200 ml of dry wine or 50 ml of spirits), or total abstaining from alcohol consumption for the study period.

Exclusion Criteria:

1. Chronic liver disease of any other aetiology.
2. Disorders of copper metabolism, and/or ceruloplasmin serum level beyond the reference value on screening.
3. Disorders of iron metabolism in the past medical history or revealed at screening.
4. Cirrhotic stage of nonalcoholic fatty liver disease (Class A-C by Child-Pugh).
5. Type I diabetes mellitus.
6. Type II diabetes mellitus, which requires regular oral hypoglycemic therapy or insulin, or the level of fasting plasma glucose> 7 mmol / l and / or glycosylated hemoglobin> 7% on screening.
7. Any severely decompensated somatic disease
8. Regular intake of the medications that are prohibited by the study protocol, or their intake within 4 weeks prior to inclusion.
9. The history of clinically significant allergic reactions.
10. Hypersensitivity to any component of the study drug and / or intolerance to any component of the study drug.
11. Bariatric surgery in less than 6 months prior to the study.
12. Pregnancy or lactation.
13. Hyperhomocysteinemia (homocysteine serum levels >15 mmol/dL for men, >12 mmol/dL for women).
14. Exacerbation of the stomach ulcer and / or duodenal ulcers and / or erosive gastritis.
15. Chronic kidney failure (stage C4-C5) and / or glomerular filtration rate <30 ml / min on screening.
16. Gout, with the need of drugs that reduce uric acid levels
17. Any of the following parameters: Hb <80 g / L, platelets <80 x 10 9 / L, WBC> 15 x 10 9 / L at screening.
18. Regular intake of more than 5 units of alcohol per week (1 unit of alcohol is equivalent to 0.5 liters of beer, 200 ml of dry wine or 50 ml of spirits) or history of alcohol addiction.
19. A significant (over 5 kg) weight loss or weight gain during the preceding 6 months prior to the study.
20. Unstable angina pectoris.
21. Myocardial infarction within 3 months before inclusion.
22. Chronic heart failure (III-IV functional class by NYHA).
23. A history of cancer, mental illness, HIV, tuberculosis, or drug addiction.
24. Mental, physical and other reasons that do not allow the patient to comply with the study procedures.
25. Any other condition which, according to the investigator's judgement, may interfere with the compliance to study procedures.
26. Participation in any other clinical trial within 3 months prior to the inclusion.
27. Employees of the research company or study site involved in the conduct of the present study, and their family members.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Proportion of responders to treatment | 102 days, including the screening period (14 days)
  The proportion of responders with non-alcoholic fatty liver disease, as demonstrated by assessment of liver function by the following laboratory findings: decrease in ALT and AST iby at least 40% from baseline, and / or reduction of GGT by at least 30% from baseline at the end of the course of treatment

SECONDARY OUTCOMES:
Severity of dyslipidemia | 102 days, including the screening period (14 days)
  The dynamics of the severity of atherogenic dyslipidemia (as demonstrated by the level of total cholesterol, triglycerides, cholesterol, low density lipoprotein (LDL), high density lipoprotein cholesterol (HDL-C)) in patients by the end of the therapeutic course in comparison with baseline findings
The insulin resistance index (HOMA-IR) | 102 days, including the screening period (14 days)
  The change of the insulin resistance index (index HOMA-IR, calculated according to the level of fasting plasma glucose, fasting insulin) in patients by the end of the treatment course in comparison with the baseline findings
Transaminases | 102 days
  Dynamics of transaminases serum levels (ALT, AST) in patients between the study visits
cholestasis markers (alkaline phosphatase, GGT) | 102 days
  Dynamics of cholestasis markers (alkaline phosphatase, GGT) in the serum of patients between study visits
Bilirubin | 102 days
  Dynamics of total bilirubin serum levels (ALT, AST) in patients between the study visits
Body mass index | 102 days
  Change of the BMI of patients at the end of the treatment course in comparison with the baseline measurements
ultrasound signs of hepatic steatosis | 102 days
  Dynamics of ultrasound signs of hepatic steatosis in patients by the end of the treatment course in comparison with the baseline

OTHER OUTCOMES:
Serum homocysteine | 102 days
  homocysteine serum level at screening and at all study visits

CONTACTS AND LOCATIONS:
Overall Officials: Igor G Nikitin, Principal Investigator — Central Clinical Hospital of the Russian Academy of Sciences; Vladimir B Grinevich, Principal Investigator — Military Medical Academy named after SM Kirov," the Russian Defense Ministry, 2nd Department and Clinic of medical postrgaduate education; Alexander V Gordienko, Principal Investigator — Military Medical Academy named after SM Kirov," the Russian Ministry of Defense, Hospital Therapeutic Department and Clinic; Vyacheslav G Morozov, Principal Investigator — Medical company "Hepatologist" Ltd.; Vladimir V Gorbakov, Principal Investigator — Company "Clinic of professor Gorbakov" Ltd.; Chavdar S Pavlov, Principal Investigator — First Moscow State Medical University named after IM Sechenov, Russian Federation Ministry of Public Health, University Clinical Hospital №2,; Michael A Osadchuk, Principal Investigator — First Moscow State Medical University named after IM Sechenov, Health Ministry of the Russian Federation, Outpatient Department; Andrew Yu Baranovsky, Principal Investigator — St. Petersburg State health care institution "City Clinical Hospital №31"; Lyudmila S Oreshko, Principal Investigator — Federal State Educational Institution of Higher Education "Northwest State Medical University named after II Mechnikov," the Ministry of Health and Social Development of the Russian Federation; Viktor D Pasechnikov, Principal Investigator — Stavropol State Medical University, Ministry of Health of the Russian Federation, Department of therapy with a course of dietetics; Maria A Livzan, Principal Investigator — Omsk State Medical Academy, Ministry of Health and Social Development of the Russian Federation, Department of faculty therapy; Yuri P Uspenskiy, Principal Investigator — St. Petersburg City Hospital of the Holy Martyr Elizabeth; David L Nepomnyashchikh, Principal Investigator — State Novosibirsk Regional Clinical Hospital; Polina M Hlyabova, Principal Investigator — Limited Liability Company "BioEk" Ltd.; Sergei L Grishaev, Principal Investigator — St. Petersburg state healthcare institution "Mariinsky Outpatient Clinic"
Locations (3):
- Russia (3):
  - Company "Clinic of professor Gorbakov" Ltd., Krasnogorsk
  - City Hospital of the Holy Martyr Elizabeth, Saint Petersburg
  - Medical Company "Hepatologist" Ltd., Samara

IPD SHARING:
Plan to Share IPD: Undecided